CLINICAL TRIAL: NCT02370927
Title: Pulse EnRiched Food and Exercise Clinical Trials (PERFECT Project): Part 2 - Acute Effects of Pulse Ingredients in Food Products on Aerobic Endurance and Substrate Oxidation During Exercise, as Well as, the Blood Glucose, Insulin, Lactate and Food Intake Response Following an Endurance Exercise Session in Adults - Study 2
Brief Title: PERFECT Project - Part 2 - Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Saskatchewan Pulse Growers (Other); Alberta Pulse Growers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: B2014:114-4
Record Dates: First submitted 2014-12-17; First posted 2015-02-25 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Prevention; Obesity Prevention
MeSH Terms: interventions — Pea Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- Control (Placebo Comparator): 100% Wheat Flour
  Interventions: Other: Control
- Cereal w/ pea protein (Experimental): Pea protein
  Interventions: Other: Pea protein
- Cereal w/ pea starch (Experimental): Pea starch
  Interventions: Other: Pea Starch
- Cereal w/ pea starch + pea fibre (Experimental): Pea starch + pea fibre: 5g
  Interventions: Other: Pea fibre + pea starch
- Cereal w/ pea protein + pea starch (Experimental): Pea protein + pea starch: 10g
  Interventions: Other: Pea protein + pea starch
- Cereal w/ pea protein + pea fibre + pea starch: (Experimental): Pea protein + pea fibre + pea starch: 20g
  Interventions: Other: Pea fibre + pea starch + pea protein

INTERVENTIONS:
Other: Control — Non pulse extruded cereal
  Arms: Control
Other: Pea protein — Pulse extruded cereal
  Arms: Cereal w/ pea protein
Other: Pea Starch — Pulse extruded cereal
  Arms: Cereal w/ pea starch
Other: Pea fibre + pea starch — Pulse extruded cereal
  Arms: Cereal w/ pea starch + pea fibre
Other: Pea protein + pea starch — Pulse extruded cereal
  Arms: Cereal w/ pea protein + pea starch
Other: Pea fibre + pea starch + pea protein — Pulse extruded cereal
  Arms: Cereal w/ pea protein + pea fibre + pea starch:

SUMMARY:
The objectives are to test the acute effects of different cereals containing pulse ingredients on: 1) aerobic endurance and substrate oxidation during exercise 2) response of blood glucose, insulin and appetite to an aerobic exercise session, and 3) food intake two hours following the exercise session. The investigators hypothesize that consumption of cereals containing pulse ingredients 60 minutes before exercise will increase aerobic endurance (lower oxygen consumption), decrease carbohydrate oxidation (greater respiratory quotient), and a reduction in lactate production during compared to the same exercise session following the ingestion of a non-pulse food. The investigators also hypothesize that consumption of cereals containing pulse ingredients will lead to lower blood glucose, insulin, appetite and food intake, suggesting lower calorie compensation, following a 60-minute aerobic exercise session compared to the same exercise session following the ingestion of a non-pulse food.

ELIGIBILITY:
Inclusion Criteria:

* Normoglycemic (<5.6 mmol/L) and normotensive (systolic blood pressure <140 mm Hg and diastolic blood pressure below < 90 mm Hg)
* Body Mass Index of 18.5-29.9 kg/m2

Exclusion Criteria:

* Restrained eaters
* Regularly skip breakfast
* Smokers
* Those on medications that may influence study outcomes or have experienced any gastrointestinal related health conditions/surgeries over the past year
* Those who are active (organized activities or athletic training at a high intensity; ≥ 150 minutes per week of moderate to vigorous physical activity)
* Those unable to walk for an hour continuously

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Plasma Glucose Concentrations | 0-240 minutes
  Measured in blood using intravenous catheter. Glucose will be determined by automated methods using Abbot Spectrum Clinical Chemistry-X Analyzer,
Food Intake | at 240 minutes
  Ad-libitum meal
Subjective Appetite | 0-240 minutes
  Motivation-to-eat Visual Analog Scale questionnaire
Exercise intensity | 60-120 minutes
  Oxygen consumption measured during exercise at 3 time points
Insulin concentrations | 0-240 minutes
  Measured in blood using intravenous catheter. and Insulin will be measured by commercially available radioimmunoassay (RIA) kits

SECONDARY OUTCOMES:
Palatability measured by Visual Analog Scale questionnaire | 5 and 260 minutes
  Food tasting
Physical comfort measured by Visual Analog Scale questionnaire | 0-240 minutes
  Contributions from energy intake
Energy/fatigue measured by Visual Analog Scale questionnaire | 0 - 240 minutes
  Estimate of energy expenditure
Heart rate | 60-120 minutes
  To monitor exercise intensity and give a measure of fatigue (cardiovascular drift)
Substrate Oxidation | 60-120 minutes
  Respiratory quotient measured during exercise at 3 time points
Lactate concentration | 60-120 minutes
  Measured before, during, and after exercise exercise at 3 time points

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, PhD, Principal Investigator — University of Manitoba, Richardson Centre for Functional Foods and Nutraceuticals
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada